CLINICAL TRIAL: NCT03248336
Title: Objective Assessment of Disparity Vergence After Treatment of Symptomatic Convergence Insufficiency (CI) in Children
Brief Title: Objective Assessment of Disparity Vergence After Treatment of Symptomatic CI in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salus University (Other)
Responsible Party: Principal Investigator, Mitchell Scheiman, Dean of Research, Salus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMS1312
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Convergence Insufficiency
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: Eligible participants received 12 weeks of office vergence/accommodative therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vision therapy group (Experimental): Twelve, 60-minute, weekly visits of office-based vergence/accommodation therapy will be administered by a trained therapist combined with procedures to practice at home (15 minutes, 5 times per week). This treatment sequence is a well-accepted approach for treatment of CI and has been successfully implemented in previous studies. Fifteen minutes of home-based therapy was prescribed to be performed 5 days per week, and compliance with home-based therapy was monitored at each visit by the therapist
  Interventions: Procedure: office-based vergence/accommodative therapy

INTERVENTIONS:
Procedure: office-based vergence/accommodative therapy — one -to-one treatment by a trained therapists. The subject is asked to perform 5-6 therapy procedures during a 60 minute therapy session. The subject is also asked to perform 15 minutes per day of home-based therapy.
  Other Names: optometric vision therapy

SUMMARY:
This study is designed to evaluate changes in objective measures of disparity vergence after office-based vergence/accommodative therapy (OBVAT) for convergence insufficiency (CI) in children 12-17 years old.

DETAILED DESCRIPTION:
30 participants with normal binocular vision and 30 with CI will be recruited for this prospective study. All participants with CI will be treated with 12 weeks of office-based vergence/accommodative therapy. The primary outcome measure will be the average peak velocity for 4° symmetrical convergence steps. Other objective outcome measures of disparity vergence will be time to peak velocity, latency, and accuracy. Changes in clinical measures [near point of convergence (NPC), positive fusional vergence at near (PFV)] and symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CI Symptom Survey score ≥ 16
* Exophoria at near at least 4 greater than at far
* Receded near point of convergence (NPC) of 6 cm break
* Insufficient positive fusional vergence (PFV) at near (i.e., failing Sheard's criterion or PFV ≤15 base-out break)
* Best-corrected distance visual acuity of 20/25 or better in each eye
* Random dot stereopsis appreciation of 500 seconds of arc or better
* Wearing appropriate refractive correction (spectacles of contact lenses) for at least 2 weeks prior to final determination of eligibility for any of the following uncorrected refractive errors (based on cycloplegic refraction within prior 12 months)
* No use of BI prism or plus add at near for 2 weeks prior to study and for duration of study

Exclusion Criteria:

* Constant strabismus at distance or near
* Esophoria of ≥ 2∆ at distance
* Vertical heterophoria ≥ 2∆ at distance or near
* ≥ 2 line interocular difference in best-corrected visual acuity
* Near point of accommodation >20 cm in either eye as measured by push-up method
* Manifest or latent nystagmus
* History of strabismus surgery or refractive surgery
* CI associated with head trauma or known disease of the brain
* Diseases known to affect accommodation, vergence, or ocular motility
* Inability to comprehend and/or perform any study-related test

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-09-02 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in average peak velocity for 4° symmetrical convergence steps after 12 weeks of therapy | After 12 weeks of therapy
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and the primary outcome measures will be the change in average peak velocity for 4° symmetrical convergence steps

SECONDARY OUTCOMES:
Change in time to peak velocity for 4° symmetrical convergence steps after 12 weeks of therapy | After 12 weeks of therapy
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in time to peak velocity for 4° symmetrical convergence steps
Change in latency for 4° symmetrical convergence steps after 12 weeks of therapy | After 12 weeks of therapy
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in latency for 4° symmetrical convergence steps
Change in accuracy for 4° symmetrical convergence steps after 12 weeks of therapy | After 12 weeks of therapy
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in accuracy for 4° symmetrical convergence steps
Change in settling time for 4° symmetrical convergence steps after 12 weeks of therapy | After 12 weeks of therapy
  The ISCAN RK-826PCI binocular tracking system (Burlington, MA) will be used used to objectively record horizontal vergence eye movements. Five parameters will be measured with this instrument and a secondary outcome measures will be the change in settling time for 4° symmetrical convergence steps
Change in the near point of convergence | After 12 weeks of therapy
  The near point of convergence will be measured using the Near Point Rule at baseline and after 12 weeks of therapy. The change in this measurement will a secondary clinical outcome measure.
Change in the positive fusional vergence | After 12 weeks of therapy
  Positive fusional vergence will be measured using a handheld target placed 40 cm from the participant and using a horizontal prism bar. Positive fusional vergence will be measured at baseline and after 12 weeks of therapy. The change in this measurement will a secondary clinical outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No